CLINICAL TRIAL: NCT05516225
Title: Phase 1 Safety Study of Human Milk Oligosaccharide Concentrate PBCLN-003 in Healthy Adult Volunteers
Brief Title: Safety Study of Human Milk Oligosaccharides in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prolacta Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 16-CLN-003
Record Dates: First submitted 2022-08-22; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PBCLN-003, 1.8 g daily in 3 divided oral doses for 7 days (Experimental)
  Interventions: Drug: PBCLN-003
- PBCLN-003, 3.6 g daily in 3 divided oral doses for 7 days (Experimental)
  Interventions: Drug: PBCLN-003
- PBCLN-003, 9 g daily in 3 divided oral doses for 7 days (Experimental)
  Interventions: Drug: PBCLN-003
- PBCLN-003, 18 g daily in 3 divided oral doses for 7 days (Experimental)
  Interventions: Drug: PBCLN-003

INTERVENTIONS:
Drug: PBCLN-003 — Human Milk Oligosaccharide Concentrate

SUMMARY:
First-in-human phase 1 study conducted in healthy adult male and female volunteers to determine the safety and tolerability of increasing doses of PBCLN-003, which are concentrated human milk oligosaccharides (HMO).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 and 24.9 kg/m2
* Age between 18 and 50 years old
* No diagnosed medical conditions
* No significant change to diet in the 2 weeks prior to enrollment
* Agreement to use contraception for female subjects

Exclusion Criteria:

* Lactose intolerance
* Pregnancy
* Lactation
* Enrollment in another clinical study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2017-02-13 (Actual); Study Completion 2017-02-13 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 28 days
  Adverse events include those reported by questionnaire or detected as an abnormality on physical examination, laboratory testing (hematology, biochemistry, urinalysis), and 12-lead electrocardiogram.

SECONDARY OUTCOMES:
Stool, saliva, and vaginal microbiome | 28 days
  16S ribosomal RNA gene sequencing and shotgun metagenomics will be performed to detect relative abundances of bacteria at the level of 97% operational taxonomic units. Alpha diversity will be measured using the Shannon index.
Serum cytokine levels | 28 days
  IL2, IL4, IL5, IL6, IL10, IL12, TNFα, IFNγ, and TGFβ measured by ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- WCCT Global, LLC, Cypress, California, United States

REFERENCES:
- [Derived] Jacobs JP, Lee ML, Rechtman DJ, Sun AK, Autran C, Niklas V. Human milk oligosaccharides modulate the intestinal microbiome of healthy adults. Sci Rep. 2023 Aug 31;13(1):14308. doi: 10.1038/s41598-023-41040-5. PMID 37652940